CLINICAL TRIAL: NCT01414803
Title: Tolerability and Efficacy of Rosuvastatin - Fenofibrate Combine Therapy in Korean Patients With Combined Hyperlipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Yangsoo Jang/Professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2008-0390
Record Dates: First submitted 2011-08-03; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Hyperlipidemia
Keywords: rosuvastatin, fenofibrate, creatine kinase, alanine aminotransferase
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rosuvastatin/fenofibrate combination (Experimental): rosuvastatin 10 mg/fenofibrate 160 mg per day
  Interventions: Drug: Lipid modification
- rosuvastatin monotherapy (Active Comparator): rosuvastatin 10 mg per day
  Interventions: Drug: Lipid modification

INTERVENTIONS:
Drug: Lipid modification — rosuvastatin 10 mg/fenofibrate 160 mg per day
  Arms: rosuvastatin/fenofibrate combination
Drug: Lipid modification — rosuvastatin 10 mg per day
  Arms: rosuvastatin monotherapy

SUMMARY:
Although the combination of statin and fenofibrate is one of the options for patients with combined hyperlipidemia, non-lipid effects of it has not been completely understood yet. In this study we compared the effects of rosuvastatin 10 mg/fenofibrate 160 mg combination and rosuvastatin 10 mg monotherapy on muscle and liver enzyme, homocysteine levels, kidney, blood glucose control, and blood cell counts.

ELIGIBILITY:
Inclusion Criteria:

* mixed hyperlipidemia: total cholesterol levels higher than 220 mg/dL, triglyceride (TG) levels between 200 and 500 mg/dL, and low-density lipoprotein (LDL)-cholesterol levels higher than 130 mg/dL after 6-week diet/life style change
* Men and women who were between 20 and 70 years of age
* Having at least one history of: coronary artery disease, cerebrovascular disease or transient ischemic attack, peripheral vascular disease, or diabetes mellitus.
* Having risk factors at least two of: age ≥45 years in male or ≥55 years in female, elevated blood pressure (systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg, or treatment of previously diagnosed hypertension), high-density lipoprotein (HDL)-cholesterol <40 mg/dL, family history of coronary artery disease at age <55 years in male or <65 years in female, central obesity (waist circumference ≥90 cm for male or ≥80 cm for female), fasting plasma glucose ≥110 mg/dL, or left ventricular hypertrophy on electrocardiogram
* Written informed consent.

Exclusion Criteria:

* pregnant or breast-feeding
* uncontrolled hypertension
* uncontrolled diabetes mellitus
* thyroid dysfunction
* serum transaminase level >2 times the upper limit of normal
* history of gall bladder disease
* chronic alcoholic
* serum creatinine level >1.5 mg/dL
* history of myopathy
* history of acute myocardial infarction or acute stroke within 3 months before the study began
* acute or chronic infection or inflammation
* history of cancer
* history of adverse events associated with test drugs.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incidence of elevation of CK>5x ULN or AST>3x ULN or ALT>3x ULN | 24 weeks after drug treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Paterson JM, Smith SM, Simpson J, Grace OC, Sosunov AA, Bell JE, Antoni FA. Characterisation of human adenylyl cyclase IX reveals inhibition by Ca(2+)/Calcineurin and differential mRNA plyadenylation. J Neurochem. 2000 Oct;75(4):1358-67. doi: 10.1046/j.1471-4159.2000.0751358.x. PMID 10987815
- [Derived] Lee SH, Cho KI, Kim JY, Ahn YK, Rha SW, Kim YJ, Choi YS, Choi SW, Jeon DW, Min PK, Choi DJ, Baek SH, Kim KS, Byun YS, Jang Y. Non-lipid effects of rosuvastatin-fenofibrate combination therapy in high-risk Asian patients with mixed hyperlipidemia. Atherosclerosis. 2012 Mar;221(1):169-75. doi: 10.1016/j.atherosclerosis.2011.12.042. Epub 2012 Jan 5. PMID 22269152